CLINICAL TRIAL: NCT04446559
Title: Effect of " Sitting in a Chair " Versus " Conventional Semi-recumbent In-bed Position " on the Oxygenation Level for ICU Non-sedated Patients
Brief Title: Sitting Position and Blood Oxygenation in ICU Patient
Acronym: FALCON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHRO-2020-03
Record Dates: First submitted 2020-06-17; First posted 2020-06-25 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: ICU Patient
Keywords: Bed Rest; Sitting Position; Intensive Care Unit; Semi-recumbent Position
MeSH Terms: interventions — Sitting Position

STUDY DESIGN:
Intervention Model Description: Once the patient is included and the randomization is made, the positioning method will be applied for only one period of 3 hours (if optimal tolerance) and arterial gasometry in relation to the main objective will only be performed on this occasion. For the rest of the stay, the patient will benefit from the usual examinations and positioning techniques in the corresponding ICU.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sitting in a chair position (Experimental): For patients randomized in the chair group, we will perform the transfer to the chair immediately after the morning arterial blood gas. The chair position will be maintained for 3 hours, if the patient shows no clinical signs of discomfort or intolerance.
  Interventions: Procedure: Sitting in chair position
- Semi-recumbent in bed position (No Intervention): The patient will benefit from conventional positioning techniques in the ICU bed. With the help of the medical monitoring software present in the wards, we will note the different nursing care given to the patient during the 3 hours following the morning arterial gasometry.

INTERVENTIONS:
Procedure: Sitting in chair position — For patients randomized in the chair group, we will perform the transfer to the chair immediately after the morning arterial blood gas. The chair position will be maintained for 3 hours, if the patient shows no clinical signs of discomfort or intolerance.
  Arms: Sitting in a chair position

SUMMARY:
The positioning of the ICU patient is a daily concern of the medical and paramedical teams. Developments in emergency medicine and sedation and analgesia techniques have made it possible to reduce patient mortality. However, considered too unstable, patients were no longer mobilized outside the bed until the complete resolution of the symptoms that led to hospitalization or surgery.

Despite encouraging results for early mobilization, bed and rest remained the most widespread positioning technique worldwide with the emergence of intensive care units, mechanical ventilation and sedation/analgesia/curarization. The result is peripheral muscular amyotrophy and respiratory muscular amyotrophy, with increased length of stay and exacerbated morbidity/mortality several years after discharge from ICU.

Numerous studies have shown the value of early mobilization of the ICU patient to preserve functional and muscular capital.

However, few studies have evaluated the value of mobilizing the ICU patient from the bed in order to improve oxygenation. The lack of mobility outside the bed causes condensation of the pulmonary parenchyma at the bases and in the dorsal region when the patient is lying down or in a prolonged semi-seated position.

In awake spontaneously ventilated patients, whether intubated on ventilatory support (Pressure Support), non-invasive ventilation (NIV) or high flow nasal oxygen therapy (HFNO), the reference position is a semi-seated patient with the head of the resuscitation bed tilted at 30°. The problem with this position in the bed is that patients tend to slide toward the foot of the bed. This migration is due to gravity or the design of the ICU bed. The end result of this migration is that the inclination indicated by the bed head inclinometer does not correspond to the actual angulation between the patient's lower limbs and trunk. The patient finds himself "compressed" in the lower abdomen, which can lead to compression of the diaphragm and thus hypoventilation in the postero-caudal regions of the lungs.

Our hypothesis is that the chair position (outside the ICU bed) allows, without modification of the ventilatory parameters, to improve the alveolar ventilation and thus the oxygenation of the arterial blood, compared to the "natural" semi-seated position in the ICU bed, in patients with spontaneous ventilation (PS/NIV/HFNO).

DETAILED DESCRIPTION:
This is a monocentric, comparative, randomized, open-label trial comparing two methods of "seated" positioning of the ICU patient, chair versus natural position in bed, on arterial blood oxygenation

1. Sitting in a Chair position For patients randomized in the chair group, we will perform the transfer to the chair immediately after the morning arterial blood gas. The chair position will be maintained for 3 hours, if the patient shows no clinical signs of discomfort or intolerance.
2. Semi-recumbent position in bed The patient will benefit from conventional positioning techniques in the ICU bed. With the help of the medical monitoring software present in the wards, we will note the different nursing care given to the patient during the 3 hours following the morning arterial gasometry.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old in intensive care unit (ICU) or surgical intensive care unit (SICU)
* Intubated and under mechanical invasive ventilation for at least 24 hours or under non-invasive ventilation for more than 12 hours a day or under continuous high-flow nasal oxygen therapy for more than 24 hours or alternating NIV/HFNO.
* Patient or next of kin who has expressed consent to participate in the study

Exclusion Criteria:

* Tracheotomized patient
* Patient with a contraindication to sitting in a chair

  * Deep vein thrombosis not effectively anticoagulated
  * Fracture or orthopaedic disorder contra indicating mobilization
  * Lung Embolism
  * Hemodynamic instability with Average Arterial Pressure < 65 mmHg or a vasopressor amine dose greater than 0.5 ug/kg/min
* Pregnant or breastfeeding woman
* Therapeutic limitation with decision of non-reintubation in case of extubation failure
* Non-affiliated or non-beneficiary patient of a social security scheme
* Person deprived of liberty by judicial or administrative decision
* Person under guardianship or curators
* Patient already included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2024-07-06 (Actual); Study Completion 2024-07-06 (Actual)

PRIMARY OUTCOMES:
Evolution of the PaO2/FiO2 ratio between arterial gasometry at the end of the night and arterial gasometry at the end of the positioning sequence. | Hour 3
  Comparison of the PaO2/FiO2 ratio between early seating out of the bed for ICU patient under spontaneous breathing (NIV/PS/HFNO) and patients in the natural in bed position.

SECONDARY OUTCOMES:
Incidence of intolerance criteria regarding the randomization group. | Hour 3
  The objective is to compare between the two groups the clinical tolerance during positioning

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume FOSSAT, Principal Investigator — CHR Orléans
Locations (1):
- CHR d'Orléans, Orléans, France

REFERENCES:
- [Background] Domanski Z, Niezabitowski K, Latawiec-Mazurkiewicz I. [Phlebography of the spermatic vein near the unpalpable testicle]. Rofo. 1980 Sep;133(3):322-4. No abstract available. German. PMID 6110624
- [Background] Castellani G, Vincenzi G, Brugnolo E. [Reliability of parapulp support in the coronal reconstruction of silver amalgam in posterior teeth]. Dent Cadmos. 1983 Jun;51(6):25-32. No abstract available. Italian. PMID 6583091